CLINICAL TRIAL: NCT01112813
Title: The Neurotrophic Effects of Lithium Carbonate Following Stroke: A Feasibility Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Li-2010
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2017-10

CONDITIONS: Stroke
Keywords: Stroke; lithium; MRI; gray matter
MeSH Terms: conditions — Stroke | interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lithium (Experimental): Lithium Carbonate, 0.4-0.8 mmol/L for 2 months
  Interventions: Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Lithium Carbonate — 0.4-0.8 mmol/L for 2 months
  Other Names: Carbolith

SUMMARY:
Stroke is the leading cause of adult disability and the third leading cause of death in Canada. Most stroke survivors live with residual impairments that diminish independence and quality of life. This may include vascular cognitive impairment (loss of ability to plan, think and reason) which can lead to dementia and loss of mental and functional independence.

The current treatment to reduce stroke induced brain tissue injury is limited to thrombolytics (clot busters), a therapy useful only if given in the first hours following stroke. One major new approach aims to reduce cell death after stroke by targeting the ongoing tissue loss initiated by the stroke. The tissue can be maintained by interfering with later neurochemical processes that are activated by stroke, potentially through activating natural substances in the brain that help survival and growth of nerve cells ("neurotrophic" factors).

The recent recognition of lithium as a neurotrophic agent has generated the first studies of lithium treatment for managing brain diseases. Clinically, lithium has now been shown to increase brain gray matter volume in bipolar patients. This effect is potentially important in stroke because gray matter loss has been implicated in the development of cognitive impairment after stroke, a result of the series of brain processes that are activated by lack of oxygen due to stroke. Our primary objective is to examine the effects of lithium on total brain gray matter volume in the post-stroke population, as measured by volumetric magnetic resonance imaging (MRI) with the hope that lithium may increase gray matter volume in post-stroke patients and lead to greater cognitive and functional rehabilitation. This study will provide valuable information on the tolerability of lithium, and its effects on clinical outcomes relevant to stroke, providing the information needed for designing a large-scale clinical trial.

DETAILED DESCRIPTION:
The recognition of lithium as a neurotrophic agent has provided a rationale for evaluation of this agent in animal models of cerebral ischemia. Numerous animal and in vitro studies have shown lithium-mediated neurotrophic effects involve mechanisms highly relevant to the post-stroke population: the induction of brain-derived neurotrophic factor (BDNF) and inhibition of abnormal activity of glycogen synthase kinase 3 (GSK-3). Lithium has consistently been shown to increase serum concentration of the neurotrophic factor, BDNF. BDNF is involved with neuronal proliferation, survival, and differentiation and it facilitates cortical reorganization and functional recovery after focal ischemia (in rats). GSK-3 is a neurotrophic intermediary. In animal and in vitro models, lithium treatment effectively reduces the severity of ischemic damage and protects against ischemic damage of central nervous system (CNS) neurons resulting from glutamate-induced cell death. Importantly, these benefits were present when lithium was given after ischemic events rather than prophylactically.

The goal of pharmacotherapy post-stroke is to enhance restoration of neurological function and limit structural degradation. Gray matter atrophy is a relevant post-stroke relevant outcome as it has been implicated in the development of vascular cognitive impairment after stroke and is a result of the series of neurochemical processes that are activated by ischemia. While the first clinical studies examining the neurotrophic effects of lithium and its effects on total gray matter volume in bipolar subjects have just emerged, this has yet to be explored in the post-stroke population. Our primary objective is to determine the tolerability of lithium following a stroke and to examine its effects on clinical outcomes including total brain gray matter volume as measured by volumetric magnetic resonance imaging (MRI).

In this feasibility study, lithium carbonate (target 0.4 to 0.8 mmol/L) will be given open-label for 60 days, to consenting patients with unilateral ischemic cortical lesions. Total gray matter volume using magnetic resonance imaging will also be measured at baseline and termination, and related to changes in clinical outcomes (standardized scales measuring cognitive, activities of daily living, motor recovery) performed at the time of the MRIs. We expect to find that post-stroke patients receiving lithium will have increases in gray matter volume, and that increase in gray matter volume will predict improvements in clinical outcomes over 60 days. In addition, since lithium has been shown to increase serum concentration of the neurotrophic factor, BDNF, we will explore the relationship between plasma BDNF concentrations and neurological and clinical outcomes.

This study will provide key information of clinical importance that will determine whether a clinical trial with lithium is desirable and feasible. Results of this project have the potential to focus the development of lithium as a new treatment strategy that would improve outcomes at both the individual and societal level.

ELIGIBILITY:
Inclusion Criteria:

* age >40 years
* male or female
* speaks and understands English
* within 12 months post-stroke

Exclusion Criteria:

* subarachnoid or intracranial hemorrhage
* severe aphasia or dysphasia
* impaired level of consciousness that would preclude neuropsychiatric testing
* significant acute medical illness that may contraindicate lithium treatment(including renal dysfunction; >106 umol/L creatinine level) affect neuropsychiatric assessments or serum BDNF results or put subject at risk from MRI procedure
* other psychiatric (exception of post-stroke depression) or neurological illnesses
* initiation of diuretic treatment
* use of antidepressant medications or initiation of antidepressant medications during the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-04; Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Increase in total brain gray matter volumes | Baseline, 2 months

SECONDARY OUTCOMES:
Cognitive tasks of the Neurological Disorders and Stroke - Canadian Stroke Network's (NINDS-CSN) 30 min. battery | Baseline, 2 months
Serum brain-derived neurotrophic factor (BDNF) levels | Baseline, 2 months
Serum lithium and creatinine levels | 1-week, 4-weeks, 8-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Krista L Lanctôt, PhD, Principal Investigator — Sunnybrook Health Sciences Centre; Nathan Herrmann, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Sun YR, Herrmann N, Scott CJM, Black SE, Swartz RH, Hopyan J, Lanctot KL. Lithium Carbonate in a Poststroke Population: Exploratory Analyses of Neuroanatomical and Cognitive Outcomes. J Clin Psychopharmacol. 2019 Jan/Feb;39(1):67-71. doi: 10.1097/JCP.0000000000000981. PMID 30566418